CLINICAL TRIAL: NCT06122779
Title: A Phase 2A, Double-blind, Randomized, Placebo-controlled, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986435/MYK-224 in Participants With Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Study to Evaluate Safety, Tolerability and Drug Levels of BMS-986435/MYK-224 in Participants With Heart Failure With Preserved Ejection Fraction (HFpEF)
Acronym: AURORA-HFpEF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV029-1001; 2023-505919-21 (EudraCT Number); U1111-1292-8451 (Other: WHO)
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
Keywords: BMS-986435; MYK-224; Pharmacokinetics; Pharmacodynamics; Safety; HFpEF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986435 (Experimental)
  Interventions: Drug: BMS-986435
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986435 — Specified dose on specified days
  Other Names: MYK-224
  Arms: BMS-986435
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and exposure-response (E-R) of BMS-986435/MYK-224 in participants with symptomatic Heart Failure with Preserved Ejection Fraction (HFpEF).

ELIGIBILITY:
Inclusion Criteria

- Adult participants with stable, symptomatic HFpEF with a normal heart pumping ability.

Exclusion Criteria

* Participants must not have a known diagnosis of obstructive or genetic hypertrophic cardiomyopathy or infiltrative/storage disorder such as cardiac amyloidosis, or any other acute or serious condition that could interfere with assessments during the study or may pose a risk to the participant.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-07-03 (Estimated); Study Completion 2026-07-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Up to approximately 24 weeks
Incidence of serious adverse events (SAEs) | Up to approximately 24 weeks
Incidence of AEs leading to treatment discontinuation | Up to approximately 20 weeks

SECONDARY OUTCOMES:
Summary of plasma concentrations of MYK-224 | Up to approximately 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (117):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Colorado Heart and Vascular - Lakewood, Lakewood, Colorado
  - Ascension St. Vincent's Riverside Hospital - PPDS, Jacksonville, Florida
  - Local Institution - 0003, Miami, Florida
  - University of Miami FL Miller School of Medicine -1120 NW 14th St, Miami, Florida
  - Local Institution - 0014, Atlanta, Georgia
  - Local Institution - 0048, Atlanta, Georgia
  - Bluhm Cardiovascular Institute of Northwestern, Chicago, Illinois
  - Chicago Medical Research, LLC - Hazel Crest, Hazel Crest, Illinois
  - Ascension Medical Group St. Vincent - Indianapolis Heart Care, Indianapolis, Indiana
  - Local Institution - 0045, Indianapolis, Indiana
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Local Institution - 0043, St Louis, Missouri
  - Local Institution - 0117, Hackensack, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - Local Institution - 0105, Brooklyn, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center - PPDS, Rochester, New York
  - Rochester General Hospital Center for Clinical Research, Rochester, New York
  - Laurelton Heart Specialist PC - MyClinical - PPDS, Rosedale, New York
  - Duke Cardiology Clinic - PPDS, Durham, North Carolina
  - Local Institution - 0058, Cincinnati, Ohio
  - Local Institution - 0041, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Local Institution - 0104, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Angiocardiac Care of Texas - PA - PPDS, Houston, Texas
  - Local Institution - 0051, Houston, Texas
  - Local Institution - 0066, Falls Church, Virginia
- Argentina (13):
  - Corporación Médica de General San Martín, Ciudad del Libertador General San Martín, Buenos Aires
  - Local Institution - 0107, Zárate, Buenos Aires
  - Local Institution - 0115, Zárate, Buenos Aires
  - Local Institution - 0090, Córdoba, Córdoba Province
  - Local Institution - 0053, Córdoba, Córdoba Province
  - Local Institution - 0073, Rosario, Santa Fe Province
  - IPR-Investigaciones en Patologías Respiratorias, San Miguel de Tucumán, Tucumán Province
  - Centro de Especialidades Médicas CEMEDIC, Buenos Aires
  - Local Institution - 0068, Buenos Aires
  - Local Institution - 0067, Buenos Aires
  - Sanatorio Duarte Quiros, Córdoba
  - Local Institution - 0069, Salta
  - Centro de Investigaciones Clínicas Del Litoral SRL, Santa Fe
- Canada (6):
  - Hamilton General Hospital, Hamilton, Ontario
  - Medicus MFC Inc., Toronto, Ontario
  - Local Institution - 0030, Toronto, Ontario
  - Local Institution - 0040, Toronto, Ontario
  - Local Institution - 0011, Montreal, Quebec
  - Local Institution - 0035, Trois-Rivières, Quebec
- China (5):
  - Peking Union Medical College Hospital - East Campus, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Henan Science and Technology University - Jinghua Campus, Luoyang, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital, Zhejiang University School of Medicine - Jiefanglu Campus, Hangzhou, Zhejiang
- Israel (8):
  - Local Institution - 0109, Jerusalem, Jerusalem
  - Local Institution - 0113, Jerusalem, Jerusalem
  - Local Institution - 0111, Beersheba
  - Local Institution - 0112, Be’er Ya‘aqov
  - Local Institution - 0108, Haifa
  - Local Institution - 0110, Petah Tikva
  - Local Institution - 0106, Rehovot
  - Local Institution - 0116, Safed
- Italy (10):
  - Local Institution - 0027, Foggia, Apulia
  - Local Institution - 0038, Foggia, Apulia
  - Local Institution - 0019, Napoli, Campania
  - Local Institution - 0023, Milan, Lombardy
  - Local Institution - 0033, Milan, Lombardy
  - IRCCS Policlinico San Donato, San Donato Milanese, Lombardy
  - Local Institution - 0050, San Donato Milanese, Lombardy
  - Local Institution - 0052, Massa, Tuscany
  - Local Institution - 0009, Bergamo
  - Local Institution - 0017, Pisa
- Japan (5):
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji-Shi, Hyōgo
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Okayama Rosai Hospital, Okayama, Okayama-ken
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki-Shi, Osaka
- Poland (7):
  - Clinical Trials UMED Sp. z o.o., Lódz, Lódzkie
  - Local Institution - 0031, Bialystok, Podlaskie Voivodeship
  - Local Institution - 0044, Bialystok, Podlaskie Voivodeship
  - Local Institution - 0020, Lublin, Woj. Lubelskie
  - Local Institution - 0049, Lublin, Woj. Lubelskie
  - Local Institution - 0006, Krakow
  - Local Institution - 0024, Oświęcim
- South Korea (10):
  - Chungnam National University Hospital, Daejeon, Daejeon Gwang'yeogsi
  - Inha University Hospital, Junggu, Incheon Gwang'yeogsi
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
- Spain (12):
  - Local Institution - 0012, L'Hospitalet de Llobregat, Barcelona
  - Local Institution - 0025, Majadahonda, Madrid
  - Local Institution - 0047, Majadahonda, Madrid
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Local Institution - 0039, El Palmar, Murcia
  - Local Institution - 0042, Málaga, Málaga
  - Local Institution - 0026, Madrid
  - Local Institution - 0034, Madrid
  - Local Institution - 0032, Málaga
  - Hospital Nuestra Señora de Valme, Seville
  - Local Institution - 0046, Seville
  - Local Institution - 0010, Valencia
- United Kingdom (10):
  - Northwick Park Hospital, Harrow, Greater London
  - North Tyneside General Hospital, North Shields, Northumberland
  - Leeds General Infirmary - PPDS, Leeds, Yorkshire
  - Local Institution - 0057, Sheffield, Yorkshire
  - Bristol Royal Infirmary, Bristol
  - Local Institution - 0097, Dundee
  - Local Institution - 0075, London
  - John Radcliffe Hospital, Oxford
  - University Hospital of North Tees, Stockton-on-Tees
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06122779.html